CLINICAL TRIAL: NCT07319455
Title: Heart Voice: Starry Journey - A Family-Centric and Acceptance and Commitment Therapy Based Digital Narrative Intervention, on Psychological Flexibility and Mental Health in Caregivers of Children With Autism Spectrum Disorder: A Randomized Controlled Trial
Brief Title: Heart Voice: Starry Journey - A Digital ACT Intervention for ASD Caregivers
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Harbin Medical University (Other)
Responsible Party: Principal Investigator, Hanping Gao, Principal Investigator, Harbin Medical University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: HMUDQ20251221001
Record Dates: First submitted 2025-12-19; First posted 2026-01-06 (Actual); Last update posted 2026-01-06 (Actual); Status verified 2025-12

CONDITIONS: Autism Spectrum Disorder
Keywords: Acceptance and Commitment Therapy; mHealth; Digital Storytelling
MeSH Terms: conditions — Autism Spectrum Disorder

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental): Participants allocated to this arm will receive access to and use the Heart Voice: Starry Journey mobile application, a digital interactive narrative intervention based on Acceptance and Commitment Therapy (ACT) and designed from a family-centric cultural perspective. The intervention period is 6 weeks. Participants are instructed to engage with the application by progressing through its core narrative chapters and completing embedded interactive exercises (e.g., metaphor-based training, perspective-shifting tasks, and values clarification activities). They will complete the program at their own pace on their personal smartphones. In addition to using the application, participants in this arm will complete all scheduled study assessments.
  Interventions: Device: ACT-Based Mobile Application Intervention
- Wait-list Control Group (No Intervention): Participants allocated to this arm will not receive the Heart Voice: Starry Journey intervention during the active trial period. They will be instructed to continue with their usual care and routines for the duration of the study. They will complete all scheduled study assessments at the same time points as the Intervention Arm. Upon completion of the final follow-up assessment for the entire trial, participants in this arm will be granted full access to the Heart Voice: Starry Journey application.

INTERVENTIONS:
Device: ACT-Based Mobile Application Intervention — This intervention is a culturally adapted, digitally delivered interactive narrative program based on Acceptance and Commitment Therapy (ACT) for primary caregivers of children with autism. Distinguishing features include its family-centric design, which integrates ACT's core processes into scenarios simulating intergenerational decision-making and social stigma. Delivered via a mobile application over 6 weeks, it employs a branching narrative where user choices affect outcomes, a dynamic perspective-shifting mechanism between family members, and interactive metaphor-based modules (e.g., "Quicksand" for acceptance). Its development was validated through a Delphi expert consensus process, specifically tailoring content to the psychosocial stressors of caregivers in family-oriented cultural contexts.
  Other Names: Heart Voice: Starry Journey
  Arms: Intervention Group

SUMMARY:
The goal of this clinical trial is to evaluate the effectiveness of the "Heart Voice: Starry Journey" program, a family-centric and Acceptance and Commitment Therapy (ACT)-based digital narrative intervention, in improving psychological flexibility and mental health among primary caregivers of children with Autism Spectrum Disorder (ASD). The main questions it aims to answer are:

1. Does the "Heart Voice: Starry Journey" intervention lead to a greater improvement in psychological flexibility among caregivers of children with ASD, compared to a control group?
2. Does the "Heart Voice: Starry Journey" intervention lead to a greater reduction in symptoms of anxiety and depression among caregivers of children with ASD, compared to a control group? Researchers will compare the intervention group (using the "Heart Voice: Starry Journey" program) with a wait-list control group (receiving usual care and access to the intervention after the trial) to see if the digital intervention is more effective.

Participants in the intervention group will:

* Use the "Heart Voice: Starry Journey" mobile application over a 6-week period, engaging with interactive stories and ACT-based exercises.
* Complete a series of online questionnaires about their psychological flexibility, anxiety, depression, and caregiver burden at the beginning of the study, immediately after the 6-week intervention, and at a follow-up time point (1 months later).

Participants in the wait-list control group will:

* Continue with their usual care routines during the study period.
* Complete the same series of online questionnaires at the same time points as the intervention group.

ELIGIBILITY:
Inclusion Criteria:

The child being cared for has been professionally diagnosed with Autism Spectrum Disorder (ASD) according to the Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition (DSM-5).

The primary caregiver of the child with ASD (parent or legal guardian). If multiple primary caregivers exist in the family, the one with the longest caregiving time will be included.

Possesses basic cognitive and literacy skills. Provides informed consent and voluntarily agrees to participate in the study.

Exclusion Criteria:

The child being cared for has comorbid serious organic diseases (e.g., epilepsy, congenital heart disease) or neurological damage.

Currently participating in other psychological intervention studies or having received structured psychological support services within the past 3 months.

The family has experienced a major negative life event (e.g., bereavement, severe financial crisis, natural disaster) within the past 6 months.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 52 (Estimated)
Dates: Start 2026-03 (Estimated); Primary Completion 2026-07 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Psychological Flexibility | 10 weeks
  Psychological flexibility was assessed using the Comprehensive Assessment of Acceptance and Commitment Therapy Processes (CompACT) questionnaire developed by Francis et al. This study employed the Chinese version translated by Fang et al. The scale consists of 23 items across three dimensions: Openness, Awareness, and Action. It uses a 7-point Likert scale ranging from "Never" to "Always," scored from 0 to 6, with higher total scores indicating a greater level of psychological flexibility.
Parental Burnout | 10 weeks
  Developed by Roskam et al. to assess parenting burnout levels. There are 23 items in the scale, which are divided into four dimensions: the sense of exhaustion of the parental role, the boredom of the parental role, the emotional alienation from the children, and the self-comparison with the previous parental role. Scores range from 23-161. Higher scores indicate higher levels of parental burnout.
Caregiver Needs and Resources | 10 weeks
  Caregiver needs and resources were assessed using the Caregiver Needs and Resources Assessment (CNRA) scale developed by Li et al. The scale consists of 36 items across two dimensions (Needs and Resources) and 12 domains, with 2 of the items being reverse-scored. It employs a 5-point Likert scale ranging from "Never" to "Extremely Much," scored from 1 to 5. Higher scores indicate more pronounced levels of the corresponding needs or resources.

SECONDARY OUTCOMES:
Autism Knowledge | 10 weeks
  Autism knowledge was assessed using the Chinese version of the Autism Stigma and Knowledge Questionnaire (ASK-Q) revised by Zhai, which is adapted from the original instrument developed by Harrison et al. This revised version excludes the "stigma" dimension and focuses solely on knowledge assessment. The scale consists of 47 items across three dimensions: Diagnosis/Symptoms, Etiology, and Intervention. It employs a dichotomous scoring method, with "Correct" answers scored as 1 point, and "Incorrect" or "Don't Know" answers scored as 0 points. The total score ranges from 0 to 47, with higher scores indicating a better understanding of autism-related knowledge.
Caregiver Burden | 10 weeks
  Caregiver burden was assessed using the Care Burden Index (CBI), originally developed by Novak et al. to evaluate the level of burden experienced by caregivers. This study employed the Chinese version translated and validated by Zhang et al. The scale consists of 24 items across five dimensions: Time-Dependence Burden, Developmental Burden, Physical Burden, Social Burden, and Emotional Burden. It uses a 5-point Likert scale ranging from "Strongly Disagree" to "Strongly Agree," scored from 1 to 5. The total score ranges from 0 to 96, with higher scores indicating a greater level of caregiver burden.
Psychological Health Status | 10 weeks
  Psychological health status was assessed using the 21-item Depression Anxiety Stress Scale (DASS-21). This study employed the simplified Chinese version revised by Gong et al. The scale consists of 21 positively scored items across three dimensions: Depression, Anxiety, and Stress. It uses a 4-point Likert scale ranging from "Did not apply to me at all" to "Applied to me very much or most of the time," scored from 0 to 3. Higher scores indicate higher levels of depression, anxiety, and stress, reflecting poorer mental health status.
Perceived Social Support | 10 weeks
  Perceived social support was measured using the Perceived Social Support Scale (PSSS) translated and revised by Jiang et al. The scale consists of 12 positively scored items across three dimensions: Family Support, Friend Support, and Other Support. It employs a 7-point Likert scale ranging from "Very Strongly Disagree" to "Very Strongly Agree," scored from 1 to 7. Higher scores indicate a higher level of perceived social support.

OTHER OUTCOMES:
Feasibility Assessment | 10 weeks
  The feasibility assessment tool was developed by the researchers based on the system content and employs a mixed-method approach combining structured scales with open-ended feedback. The quantitative component uses a 7-point Likert scale to measure participants' overall satisfaction with the program. Additionally, subjective open-ended questions are included to gather qualitative feedback. Core prompts include: "Which part of the story impressed you the most, and why?" "What was the most helpful component of the program?" "What specific support did you gain from using the system?" and "What changes have you noticed in yourself after using the system?" Finally, an open-ended text box is provided to collect participants' overall experiences, suggestions for improvement, and any additional comments.

CONTACTS AND LOCATIONS:
Locations (1):
- Harbin Medical University, Daqing Campus, Daqing, Heilongjiang, China

IPD SHARING:
Plan to Share IPD: No